CLINICAL TRIAL: NCT04943419
Title: Myeloid-derived Suppressor Cells in Colorectal Cancer: Influence on Postoperative Complications and Neoadjuvant Treatment
Brief Title: Myeloid-derived Suppressor Cells in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, Ph D, Principal Investigator, Jagiellonian University
Other Study IDs: Colorectal MDSC
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Suppression; Complication,Postoperative; Radiotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer: Patients with colorectal cancer qualified for elective operations.
  Interventions: Diagnostic Test: Level of Myeloid-Derived Suppressor Cells

INTERVENTIONS:
Diagnostic Test: Level of Myeloid-Derived Suppressor Cells — Establishing of levels of all MDSC, PMNMDSC, MMDSC, EMDSC, M/PMN MDSC ratio on the day before operation.

SUMMARY:
The aim of the study is to evaluate whether the preoperative level of myeloid-derived suppressor cells is associated with postoperative complications classified by Clavien-Dindo categories. Levels of all MDSC, polymorphonuclear MDSC (PMNMDSC), monocytic MDSC (MMDSC), early-stage MDSC (EMDSC) and monocytic to polymorphonuclear MDSC ratio (M/PMN MDCS) were established and compared in patients with postoperative complications, severe postoperative complications (>= IIIA according to Clavien-Dindo) and severe septic complications.

DETAILED DESCRIPTION:
Levels of all MDSC, polymorphonuclear MDSC (PMNMDSC), monocytic MDSC (MMDSC), early-stage MDSC (EMDSC) and monocytic to polymorphonuclear MDSC ratio (M/PMN MDCS) were established and compared in patients with and without postoperative complications. Then subgroup analysis was performed to compare levels of MDSC in patients with severe postoperative complications (>= IIIA according to Clavien-Dindo) and those without severe complications. Another subgroup analysis will be performed for patients with severe septic complications that are defined as severe complications with accompanying infection. Levels of MDSC will be compared by means of U Mann Whitney test as their distribution is not normal. After above mentioned analyses it will be possible to evaluate the role of MDSC in patients with colorectal cancer in terms of postoperative complications. Additional analyse will be performed to compare levels of MDSC in patients who underwent neoadjuvant treatment (radiotherapy or chemoradiotherapy).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* colorectal cancer confirmed by histological examination of biopsy specimen
* elective operation
* signed informed consent

Exclusion Criteria:

* Age < 18
* Pregnancy or lactation
* Emergency operation
* General condition that precludes understanding and signing of the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically-confirmed colorectal cancer who undergo elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Level of MDSC in patients with postoperative complications | 30 days
  Level of all MDSC, polymorphonuclear MDSC (PNMMDSC), monocytic MDSC ( MMDSC), early-stage MDSC (EMDSC) and monocytic to polymorphonuclear MDSC ratio (M/PMNMDSC) in patients with postoperative complications

SECONDARY OUTCOMES:
Level of MDSC in patients with severe postoperative complications | 30 days
  Level of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio in patients with severe postoperative complications (Clavien-Dindo>= IIIA)
Level of MDSC in patients with severe septic postoperative complications | 30 days
  Level of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio in patients with severe postoperative complications (Clavien-Dindo>= IIIA) with infection
Level of MDSC in patients after neoadjuvant therapy | 1 day before surgery
  Level of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio in patients after neoadjuvant treatment
Level of MDSC in patients with T2-T4 tumours after neoadjuvant treatment | 1 day before surgery
  Level of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio in patients with tumours T2-T4 after neoadjuvant treatment
Level of MDSC measured in the specimen | 1 day
  evel of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio measured in the specimen after resection
Level of MDSC in patients with left and right sided tumours | 1 day
  evel of all MDSC, PNMMDSC, MMDSC, EMDSC and M/PMNMDSC ratio measured in patients with left-sided and right-sided colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Pach, Ph.D., Principal Investigator — Jagiellonian University
Locations (1):
- 1st Department of General Surgery, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rogala J, Sieminska I, Baran J, Rubinkiewicz M, Zybaczynska J, Szczepanik AM, Pach R. Myeloid-Derived Suppressor Cells May Predict the Occurrence of Postoperative Complications in Colorectal Cancer Patients-a Pilot Study. J Gastrointest Surg. 2022 Nov;26(11):2354-2357. doi: 10.1007/s11605-022-05364-3. Epub 2022 Jun 1. No abstract available. PMID 35650461